CLINICAL TRIAL: NCT05285319
Title: Phase II Randomized Control Trial Comparing Radical Hypofractionated Radiotherapy to Prostate Only VS Prostate And Pelvic Lymph Nodes in Intermediate And High Risk Prostate Cancer
Brief Title: Trial Comparing Radical Radiotherapy to Prostate Only VS Prostate And Pelvic Lymph Nodes in Intermediate And High Risk Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelhamid, Assistant Lecturer Of Radiation Oncology - National Cancer Institute, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RO2002-30906
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Intermediate Risk Prostate Cancer; High Risk Prostate Cancer; Hypofractionated Radiotherapy; Pelvic Lymph Node Irradiation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase II prospective randomized trial with 2 arms:
  * Prostate Only (Arm A)
    o Hypofractionated Intensity modulated radiotherapy (IMRT) to the prostate only to dose of 60Gy/20fractions (3 Gy per fraction)
  * Prostate & Pelvic Lymph Nodes (Arm B)
    * Hypofractionated Intensity modulated radiotherapy (IMRT) with elective pelvic nodes irradiation up to 44Gy/20 fractions (2.2 Gy per fraction) with a Simultaneous Integrated Boost (SIB) to the prostate to dose of 60Gy/20fractions (3 Gy per fraction)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate Only (Arm A) (Experimental): Hypofractionated Intensity modulated radiotherapy (IMRT) to the prostate only to a dose of 60Gy/20fractions (3 Gy per fraction)
  Interventions: Radiation: Prostate Only Radiation
- Prostate and Pelvic Lymph Nodes (Arm B) (Experimental): Hypofractionated Intensity modulated radiotherapy (IMRT) with elective pelvic nodes irradiation up to 44Gy/20 fractions (2.2 Gy per fraction) with a Simultaneous Integrated Boost (SIB) to the prostate to a dose of 60Gy/20fractions (3 Gy per fraction)
  Interventions: Radiation: Prostate and Pelvic Lymph Node Radiation

INTERVENTIONS:
Radiation: Prostate Only Radiation — Prostate Only Radiation for Intermediate and High Risk Prostate cancer
  Arms: Prostate Only (Arm A)
Radiation: Prostate and Pelvic Lymph Node Radiation — Prostate and Pelvic Lymph Node Radiation for Intermediate and High Risk Prostate cancer
  Arms: Prostate and Pelvic Lymph Nodes (Arm B)

SUMMARY:
This phase II randomized controlled study aims to compare the treatment results of intermediate and high risk prostate cancer patients treated with hormonal therapy and radical radiotherapy with or without pelvic lymph nodes in NCI- Cairo University.

DETAILED DESCRIPTION:
Study Design :

Phase II prospective randomized trial with 2 arms • Prostate Only (Arm A)

Hypofractionated Intensity modulated radiotherapy (IMRT) to the prostate only to dose of 60Gy/20fractions (3 Gy per fraction)

• Prostate & Pelvic Lymph Nodes (Arm B)

Hypofractionated Intensity modulated radiotherapy (IMRT) with elective pelvic nodes irradiation up to 44Gy/20 fractions (2.2 Gy per fraction) with a Simultaneous Integrated Boost (SIB) to the prostate to dose of 60Gy/20fractions (3 Gy per fraction)

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven prostatic adenocarcinoma.
* Risk stratification from intermediate to very high risk will be included according to NCCN guide lines September 5, 2019 version 4.2019:

  * Intermediate risk: T2b or T2c and/or GS =7 and/or PSA >10-20. Both the favorable intermediate (1 intermediate risk factor (IRF) and Grade Group 1 or 2 and <50% biopsy core positive) and unfavorable intermediate risk (2 or 3 IRFs and/or Grade Group 3 and/or ≥50% biopsy cores positive) will be included.
  * High risk: T3a or PSA >20 or Grade Group 4 or 5, not very high risk.
  * Very high risk: T3b-4, primary gleason pattern 5 OR >4 cores with grade group 4 or 5
* N stage: N0
* M Stage: M0
* Performance Status: PS 0-2

Exclusion Criteria:

* Low risk prostate cancer
* Histologies other than adenocarcinoma
* Patients with significant comorbidities might affect treatment completion and follow up
* Previously received pelvic radiotherapy
* Patients with metastatic disease
* Poor performance status (PS ≥ 3)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 90 days post the end of radiation therapy
  Compare Acute toxicity between the 2 arms using Radiation Therapy Oncology Group (RTOG) acute morbidity scoring criteria.
Local Control | 1 year
  Compare Local control (LC) with minimum follow up of 1 year in both groups

SECONDARY OUTCOMES:
Biochemical free survivals (BFS) | 1 year
  Biochemical free survivals (BFS) with minimum follow up of 1 year in both groups.
Late toxicity | 1 year
  Compare Late toxicity (using RTOG/EORTC Late Radiation Toxicity Scale)
Overall survival (OS) | 1 year
  Compare overall survival in the study population

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided